CLINICAL TRIAL: NCT06240897
Title: Exploring the Feasibility of Digital Intervention Games as a Diagnostic and Management Tool for Delirium at SGH Inpatient Wards
Brief Title: CURATE.Dtx as a Diagnostic and Management Tool for Delirium
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Digital Medicine (WisDM) (Other)
Collaborators: Singapore General Hospital (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: WisDM
Record Dates: First submitted 2023-10-19; First posted 2024-02-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-01

CONDITIONS: Delirium
Keywords: digital health; digital diagnostic
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital games (Experimental): Each CURATE.DTx session will be 12 minutes long. The game will be played by each participant via a study-provided tablet. During first session prior to commencing data collection, a trained trial team member will explain in detail how to play the game-based multitasking intervention. The session will require 12 minutes of gameplay for a minimum of three days and up to five days for a total duration of hospitalisation. Participants will also be encouraged to play an optional digital game that is designed to help with their emotional and cognitive health.
  Interventions: Device: CURATE.Dtx; Device: Optional games

INTERVENTIONS:
Device: CURATE.Dtx — CURATE.Dtx is a self-guided digital multitasking game that involves a combination of four subtasks played simultaneously, targeting different cognitive domains.
  Other Names: Delirium Screening Tool
Device: Optional games — The patient will first be asked how he/she feels and what they have done that day. The patient then selects a digital local pet (dog, cat, bird) and can customize its appearance, name and background location. The player can interact with their pet via several actions such as feed, bathe, train and accessorize. Playing with digital pets can help reduce stress and anxiety in the elderly. It can be a positive distraction in alleviating the elderly's worries and discomforts. In order to purchase accessories for their digital pet, they are encouraged to play short games that include Grocery Snap, Down Memory Lane and Pet Escape. These games are aimed at improving memory and reduce cognitive decline.

SUMMARY:
Inpatient delirium incidence is widely documented in international and local studies, however, there is no viable and labour-free delirium detection and management tool. CURATE.DTx is our tablet ready, multi-tasking serious game, that leverage a small data artificial intelligence-derived platform that can dynamically personalise cognitive training by modifying the game intensity. The main aims of this study are to explore the feasibility and usability of this new digital tool to aid in the delirium screening and management of at-risk delirium hospitalized patients.

DETAILED DESCRIPTION:
Delirium is a neurobehavioral syndrome caused by the acute and transient impairment of brain activity. The clinical context usually involves a vulnerable patient, susceptible to predisposing factors, such as clinical illness, cognitive and sensory deficits, with precipitating factors occurring during the period of hospitalization. Although widely documented in international and local studies, there is no viable and labour-free delirium detection tool. CURATE.DTx is our tablet ready, multi-tasking serious game, that leverage a small data artificial intelligence-derived platform that can dynamically personalise cognitive training by modifying the game intensity.

This is a single-centre, single-arm prospective cohort feasibility study. Hospitalised adults >65years old will be invited to trial the digital cognitive games. Patient experience and usability will be assessed at the end of the intervention through surveying methods. Acceptability, demand, implementation, practicality and limited accuracy testing will be assessed.

The investigators will recruit 25-50 inpatients (>65 years old adults) from the medical wards in SGH from November 2023 to Jan 2024.

Potential participants will be approached by the SGH team in person to provide more information about the study. Participants will be screened by the SGH research team for eligibility at initial contact.

Eligible participants will be invited to complete a daily cognitive evaluation session consisting of a cognitive training game session, followed by a 4 'A's Test - a well-validated bedside tool, which helps practitioners detect delirium in day-to-day practice, as well as an MMSE test as an additional measure. CURATE.DTx is a self-guided digital game-based multitasking intervention that involves a combination of four subtasks played simultaneously. The game will be played by each participant via a study-provided tablet. During first session prior to commencing data collection, a trained trial team member will explain in detail how to play the game-based multitasking intervention. The session will require 12 minutes of gameplay for a minimum of three days and up to five days for a total duration of hospitalisation. Participants will also be encouraged to play an optional digital game that is designed to help with their emotional and cognitive health. Deidentified game play data will be recorded.

Upon completing the game sessions, a survey will be administered to gather patients experience whilst using the digital tool as well as feedback on the interaction with the interface itself.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the medical ward in SGH
* Age >=65 years old
* Patients with a life expectancy of at least 1 month

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients physically incapable of using computer tablets (either due to vision loss or dominant hand weakness)
* Patients who cannot understand spoken the English language.
* Patients who are unable to give informed consent.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient Acceptability | 30 minutes
  Patient survey on acceptability of CURATE.DTx and other digital games distributed prior to discharge or at the end of 5 days
Trial Team Members Acceptability | 30 minutes
  Trial team members survey on acceptability of CURATE.DTx and other digital games distributed at the end of the trial
Demand | Throughout trial completion,up to 1 year
  Data collected during patient recruitment and throughout trial completion: a) Uptake : Percentage of successfully recruited patients from all patients approached and eligible for the study; b) Retention: Percentage of patients that complete the trial from all successfully recruited patients; c) Adherence: Percentage of completed sessions by patients at indicated timepoints
Implementation | Throughout trial completion, up to 1 year
  Data collected throughout trial completion: a) Success of CURATE.DTx execution: Number of CURATE.DTx sessions successfully performed within this setting;
Practicality | 30 minutes
  Trial team members survey on practicality of CURATE.DTx and other games distributed at the end of the trial: a) Practicality: Trial team perception of the ability of patients to carry out the activities and their potential impact; b) Logistical feasibility: Logistical considerations with current trial protocol that would need to be addressed or accounted for a future RCT

SECONDARY OUTCOMES:
Usability | 30 minutes
  Patient survey distributed prior to discharge or at the end of 5 days on usability of CURATE.DTx

CONTACTS AND LOCATIONS:
Overall Officials: Dean Ho, PhD, Principal Investigator — The Institute for Digital Medicine (WisDM); Esther M Fan Peijin, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kee, Theodore & Weiyan, Chee & Blasiak, Agata & Chong, Jordan & Chen, Jonna & Yeo, B.T. Thomas & Ho, Dean & Asplund, Christopher. (2019). Harnessing CURATE.AI as a Digital Therapeutics Platform by Identifying N-of-1 Learning Trajectory Profiles. Advanced Therapeutics. 2. 1900023. 10.1002/adtp.201900023
- [Background] Chin YC, Koh GC, Tay YK, Tan CH, Merchant RA. Underdiagnosis of delirium on admission and prediction of patients who will develop delirium during their inpatient stay: a pilot study. Singapore Med J. 2016 Jan;57(1):18-21. doi: 10.11622/smedj.2016007. PMID 26831312

DOCUMENTS (1):
  • Informed Consent Form (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT06240897/ICF_000.pdf